CLINICAL TRIAL: NCT01936467
Title: Comparison of Two Needle Aspiration Techniques for Endoscopic Ultrasound-guided
Brief Title: Comparison of Two Needle Aspiration Techniques for Endoscopic Ultrasound-guided Fine Needle Aspiration (EUS-FNA) in Solid Pancreatic Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Mouen Khashab, Assistant Professor of Medicine; Director of Therapeutic Endoscopy, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NA_00079301
Record Dates: First submitted 2013-08-29; First posted 2013-09-06 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Solid Lesions; Pancreatic Mass
Keywords: Pancreatic solid lesions; Pancreatic mass; Pancreatic cancer; Endoscopic Ultrasound; EUS; Fine needle aspiration; FNA; EUS-FNA
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard suction (Experimental): These are patients who will have endoscopic ultrasound-guided fine needle aspiration using the standard suction FNA technique: 15 to-and-fro movements within the lesion will be performed with use of 10cc suction syringe.
  Interventions: Device: Standard technique EUS-FNA
- Capillary suction (Experimental): These are patients who will have endoscopic ultrasound-guided fine needle aspiration using the capillary suction FNA technique: 15 to-and-fro movements within the lesion will be performed with simultaneous minimal negative pressure provided by pulling the needle stylet slowly and continuously.
  Interventions: Device: Capillary suction technique for EUS FNA

INTERVENTIONS:
Device: Standard technique EUS-FNA — Standard suction Endoscopic Ultrasound- Fine Needle Aspiration (EUS-FNA) technique using the 22-gauge (Expect needle; Boston Scientific) needle: 15 to-and-fro movements within the lesion will be performed with use of 10cc suction syringe.
  Arms: Standard suction
Device: Capillary suction technique for EUS FNA — Capillary suction Endoscopic Ultrasound- Fine Needle Aspiration (EUS-FNA) technique using the 22-gauge (Expect needle; Boston Scientific) needle: 15 to-and-fro movements within the lesion will be performed with simultaneous minimal negative pressure provided by pulling the needle stylet slowly and continuously
  Arms: Capillary suction

SUMMARY:
The aim of this study is to compare Endoscopic Ultrasound and Fine Needle Aspirate with a standard 22-gauge needle using either "standard-suction" or "capillary suction" methods for solid pancreatic lesions. Investigators hope to discover the best technique for obtaining diagnostic material when patients with a pancreatic mass undergo endoscopic ultrasound and fine needle aspirate procedure.

There are currently several techniques for obtaining tissue during endoscopic ultrasound and fine needle aspirate. The procedure will be performed by either the capillary suction technique or no suction technique.

ELIGIBILITY:
Inclusion Criteria:

- In-patients and out-patients between the age of 18years and 90 years with pancreatic masses presenting for EUS-FNA

Exclusion Criteria:

* Uncorrectable coagulopathy (INR > 1.5)
* Uncorrectable thrombocytopenia (platelet < 50,000)
* Uncooperative patients
* Pregnant women (women of childbearing age will undergo urine pregnancy testing, which is routine for all endoscopic procedures)
* Refusal to consent form
* Cystic lesions
* Inaccessible lesions to EUS

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mouen A Khashab, MD, Principal Investigator — Johns Hopkins Univeristy
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland

REFERENCES:
- [Derived] Saxena P, El Zein M, Stevens T, Abdelgelil A, Besharati S, Messallam A, Kumbhari V, Azola A, Brainard J, Shin EJ, Lennon AM, Canto MI, Singh VK, Khashab MA. Stylet slow-pull versus standard suction for endoscopic ultrasound-guided fine-needle aspiration of solid pancreatic lesions: a multicenter randomized trial. Endoscopy. 2018 May;50(5):497-504. doi: 10.1055/s-0043-122381. Epub 2017 Dec 22. PMID 29272906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between September 2013 and December 2014 in two tertiary academic centers
Pre-assignment Details: Patients were excluded from the study because a predominantly cystic lesion was found; the lack of an appreciable mass at EUS, unavailable on-site pathology and respiratory distress precluding completion of the examination
Groups:
- Suction Technique: These are patients who will have endoscopic ultrasound-guided fine needle aspiration using the standard suction FNA technique: 15 to-and-fro movements within the lesion will be performed with use of 10cc suction syringe.
  Standard technique EUS-FNA: Standard suction Endoscopic Ultrasound- Fine Needle Aspiration (EUS-FNA) technique using the 22-gauge (Expect needle; Boston Scientific) needle: 15 to-and-fro movements within the lesion will be performed with use of 10cc suction syringe.
- Capillary Technique: These are patients who will have endoscopic ultrasound-guided fine needle aspiration using the capillary suction FNA technique: 15 to-and-fro movements within the lesion will be performed with simultaneous minimal negative pressure provided by pulling the needle stylet slowly and continuously.
  Capillary suction technique for EUS FNA: Capillary suction Endoscopic Ultrasound- Fine Needle Aspiration (EUS-FNA) technique using the 22-gauge (Expect needle; Boston Scientific) needle: 15 to-and-fro movements within the lesion will be performed with simultaneous minimal negative pressure provided by pulling the needle stylet slowly and continuously
Period: Overall Study
Arm/Group | Suction Technique | Capillary Technique
Started | 60 | 61
Completed | 60 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suction Technique | Capillary Technique | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (13.8) | 64.2 (13.8) | 64.15 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 32 | 38 | 70
Prior History [Number; unit: participants]
  Chronic Pancreatitis | 3 | 2 | 5
  Chemotherapy | 3 | 1 | 4
  Radiation therapy | 3 | 3 | 6
Prior non-diagnostic FNA [Number; unit: participants] | 7 | 8 | 15
Antiplatelet therapy [Number; unit: participants] | 6 | 14 | 20
Pancreatic mass Location [Number; unit: participants]
  Uncinate/Head | 31 | 42 | 73
  Neck | 6 | 1 | 7
  Body | 14 | 13 | 27
  Tail | 9 | 5 | 14
Pancreatic mass size [Mean (Standard Deviation); unit: Centimeter] | 2.86 (1.23) | 3.2 (1.63) | 3.03 (1.43)
Echogeicity of the lesion [Number; unit: participants]
  Hypoecho | 52 | 55 | 107
  Isoecho | 7 | 6 | 13
  Hyperecho | 1 | 0 | 1
Cystic Component [Number; unit: mass] | 12 | 10 | 22
Vascular involvement [Number; unit: mass]
  Arterial | 28 | 21 | 49
  Venous | 28 | 32 | 60
  Arterial and Venous | 19 | 14 | 33
EUS features of chronic pancreatitis [Number; unit: participants] | 11 | 7 | 18
Biliary stent present [Number; unit: participants] — Number of patients having biliary stent at the time of EUS-FNA
  participants
    Metal stent | 1 | 5 | 6
    Plastic stent | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield of Capillary Technique
Description: Diagnostic yield is defined as percentage of specimens in which diagnostic material is obtained.
Time Frame: up to 6 months
Measure: Number; unit: percentage of specimen
Arm/Group | Capillary Technique
Number analyzed (Participants) | 61
percentage of specimen | 75.4

2. Primary Outcome: Diagnostic Yield of Standard Technique
Description: Diagnostic yield is defined as percentage of specimens in which diagnostic material is obtained.
Time Frame: up to 6 months
Measure: Number; unit: percentage of specimen
Groups:
- Standard Technique: These are patients who will have endoscopic ultrasound-guided fine needle aspiration using the standard suction FNA technique: 15 to-and-fro movements within the lesion will be performed with use of 10cc suction syringe.
  Standard technique EUS-FNA: Standard suction Endoscopic Ultrasound- Fine Needle Aspiration (EUS-FNA) technique using the 22-gauge (Expect needle; Boston Scientific) needle: 15 to-and-fro movements within the lesion will be performed with use of 10cc suction syringe.
Arm/Group | Standard Technique
Number analyzed (Participants) | 60
percentage of specimen | 65

3. Primary Outcome: Sensitivity of EUS-FNA With Capillary Technique
Description: Sensitivity of the EUS-FNA with Capillary technique
Time Frame: 6 months
Population: The discrepancy between the number of analyzed patients and the number of patients in the Participant Flow section is due to the fact that calculation of sensitivity was done based on the Per Protocol analysis.
Measure: Number; unit: participants
Groups:
- Patients With Positive Gold Standard: gold standard is defined as follows: for resectable cases, surgical histology was considered the gold standard. For unresectable or benign cases, positive cytology (with compatible clinical outcome) at 6-month follow-up was considered gold standard. Negative cytology was confirmed with clinical data and/or imaging at 6 month follow-up.
- Patients With Negative Gold Standard: These are patients who will have endoscopic ultrasound-guided fine needle aspiration using the standard suction FNA technique: 15 to-and-fro movements within the lesion will be performed with use of 10cc suction syringe.
  Standard technique EUS-FNA: Standard suction Endoscopic Ultrasound- Fine Needle Aspiration (EUS-FNA) technique using the 22-gauge (Expect needle; Boston Scientific) needle: 15 to-and-fro movements within the lesion will be performed with use of 10cc suction syringe.
Arm/Group | Patients With Positive Gold Standard | Patients With Negative Gold Standard
Number analyzed (Participants) | 48 | 4
participants
  Positive EUS-FNA | 45 | 0
  Negative EUS-FNA | 3 | 4
Statistical Analysis 1: Comparison: Patients With Positive Gold Standard vs Patients With Negative Gold Standard; Test type: Other; Sensitivity = 93.7
Statistical Analysis 2: Comparison: Patients With Positive Gold Standard vs Patients With Negative Gold Standard; Test type: Other; Specificity = 100

4. Primary Outcome: Sensitivity of EUS-FNA With StandardTechnique
Description: Sensitivity of the EUS-FNA with Capillary technique
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Patients With Positive Gold Standard | Patients With Negative Gold Standard
Number analyzed (Participants) | 44 | 0
Participants
  Positive EUS-FNA | 39 |
  Negative EUS-FNA | 5 |
Statistical Analysis 1: Comparison: Patients With Positive Gold Standard vs Patients With Negative Gold Standard; Test type: Other; Sensitivity = 88.6
Statistical Analysis 2: Comparison: Patients With Positive Gold Standard vs Patients With Negative Gold Standard; Test type: Other; Specificity = 100

5. Primary Outcome: Sensitivity of EUS-FNA
Description: Comparison of EUS-FNA sensitivity using Capillary technique versus Standard technique for pancreatic solid lesions
Time Frame: 6 months
Population: as for outcome 3
Measure: Number; unit: percentage of positive gold standard
Arm/Group | Suction Technique | Capillary Technique
Number analyzed (Participants) | 44 | 52
percentage of positive gold standard | 88.6 | 93.7
Statistical Analysis 1: Comparison: Suction Technique vs Capillary Technique; Test type: Other; p = 0.47, Chi-squared

6. Secondary Outcome: First Pass Diagnostic Rate
Description: The rate of aquiring diagnostic pancreatic mass tissue with first FNA pass
Time Frame: immediate
Measure: Number; unit: participants
Arm/Group | Suction Technique | Capillary Technique
Number analyzed (Participants) | 60 | 61
participants | 23 | 26
Statistical Analysis 1: Comparison: Suction Technique vs Capillary Technique; Test type: Superiority or Other; p = 0.71, Chi-squared

7. Secondary Outcome: Acquisition of Core Tissue
Description: The rate of acquiring core tissue of the pancreatic mass through EUS-FNA
Time Frame: immediate
Measure: Number; unit: participants
Arm/Group | Suction Technique | Capillary Technique
Number analyzed (Participants) | 60 | 61
participants | 28 | 37
Statistical Analysis 1: Comparison: Suction Technique vs Capillary Technique; Test type: Superiority or Other; p = 0.15, Chi-squared

8. Secondary Outcome: Diagnostic Accuracy of EUS-FNA
Description: The proportion of subjects without the disease with negative EUS-FNA in total of subjects without the disease
Time Frame: 6 months
Measure: Number; unit: percent accurate
Arm/Group | Suction Technique | Capillary Technique
Number analyzed (Participants) | 60 | 61
percent accurate | 88 | 93.8
Statistical Analysis 1: Comparison: Suction Technique vs Capillary Technique; Test type: Superiority or Other; p = 0.46, Chi-squared

ADVERSE EVENTS:
Arm/Group | Suction Technique | Capillary Technique
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 0/60 | 0/61

LIMITATIONS AND CAVEATS:
The endosonographers were not blinded to the procedure technique. A small possibility that cytotechnicians may have witnessed the technique. Cellularity of the specimens were not quantified. A 6 months follow-up may not detect all false negatives

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No